CLINICAL TRIAL: NCT04159974
Title: A Phase II Trial to Evaluate Safety and Efficacy of Adding Durvalumab (MEDI4736) to Standard Neoadjuvant Radiochemotherapy and of Adjuvant Durvalumab +/- Tremelimumab in Locally Advanced Esophageal Adenocarcinoma and to Evaluate Biomarkers Predictive for Response to Immune Checkpoint Inhibition
Brief Title: RICE: Radio-Immuno-Chemotherapy of Cancer of the Esophagus
Acronym: RICE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cologne (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Thomas Zander, Principal Investigator, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNI-Koeln-3571; DRKS00015218 (Registry Identifier: DRKS); 2018-003048-22 (EudraCT Number)
Record Dates: First submitted 2019-10-23; First posted 2019-11-12 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-05

CONDITIONS: Esophageal Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durvalumab (Experimental): Treatment arm A will receive durvalumab IV in a dosage of 1500mg every four weeks for 12 months as mono therapy.
  Interventions: Drug: Durvalumab 50 MG/ML
- Durvalumab + Tremelimumab (Experimental): Treatment arm B receives durvalumab in a dosage of 1500mg every 4 weeks (-3/+7 days) for 12 months post-surgery. In addition these patients receive tremelimumab IV in a fixed dose of 75mg for the first four months on day 1; 29; 57; 85 (-3/+7).
  Interventions: Drug: Durvalumab 50 MG/ML; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab 50 MG/ML — IV Infusion
Drug: Tremelimumab — IV Infusion, Combination with Durvalumab
  Arms: Durvalumab + Tremelimumab

SUMMARY:
A phase II trial to evaluate safety and efficacy of adding durvalumab (MEDI4736) to standard neoadjuvant radiochemotherapy and of adjuvant durvalumab +/- tremelimumab in locally advanced esophageal adenocarcinoma and to evaluate biomarkers predictive for response to immune checkpoint inhibition

DETAILED DESCRIPTION:
Short Study Title: RICE - Radio-Immuno-Chemotherapy of Cancer of the Esophagus

Study Phase: Phase II

Research hypothesis: The investigators aim at evaluating if (I) esophageal cancer is susceptible to immunotherapeutic approaches based on interference with the PD1 / PDL1 axis, if (II) treatment of locally advanced tumors by immunotherapeutic approaches increases cure rate and if (III) combination with radiotherapy is feasible and increases anti-tumor immunity.

Primary Objectives: The primary objective is to evaluate safety and efficacy (measured by an increase of pathological complete response rate from 20% to 35%) of the fully human monoclonal IgG1 antibody durvalumab targeting the programmed death-ligand 1 (PD-L1) in combination with neoadjuvant radiochemotherapy, followed by surgery for locally advanced esophageal cancer and cancer of the gastric esophageal junction (GEJ).

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent

  1. Study participants must have signed and dated an IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal study participant care.
  2. Study participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
* Target Population

  1. Histologically confirmed, resectable adenocarcinoma of the esophagus or cardia/gastric esophageal junction (uT3, cNx, cM0), with the following specifications:
  1. Medical and technical operability, according to the techniques described in Section 2.1.3.2.
  2. No preceding cytotoxic or targeted therapy
  3. No prior partial or complete tumor resection
* Male or female patients ≥ 18 years of age at time of study entry
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Life expectancy of at least 12 months
* Study participants must be willing to undergo at least 2 biopsies (baseline and after neoadjuvant treatment and optional in progression)
* Adequate normal organ and marrow function as defined below. Screening laboratory values must meet the following criteria and should be obtained within 28 days prior to registration WBC ≥ 1500/μL Neutrophils ≥ 1000/μL Platelets ≥ 75 x103/μL Hemoglobin > 9.0 g/dL Serum creatinine ≤ 1.5 x institutional ULN or calculated creatinine clearance (CrCl) ≥ 40 mL/min (Cockcroft-Gault)

Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

Females:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

AST/ALT (SGOT/SGPT) ≤ 2,5 x institutional ULN Total Bilirubin ≤ 1.5 x institutional ULN (except study participants with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

* Body weight > 30kg
* Reproductive Status Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception and must agree to use adequate method to avoid pregnancy for 5 months (30 days plus the time required for durvalumab to undergo five half-lives) after the last dose of study drug.

Appropriate methods of contraception are:

* female sterilization or tubal ligation (at least 6 weeks prior to the start of the study treatment),
* male sterilization (at least 6 months prior to the start of the study treatment) and/or
* a combination of a hormonal method of contraception with a barrier method or/and
* an intrauterine device or system

  * Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of β-HCG) within one until two weeks prior to the start of durvalumab at time of neoadjuvant treatment and after surgery before starting adjuvant treatment.
  * Women will be not be considered to be of childbearing potential if they are post-menopausal and/or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy). To be considered post-menopausal the appropriate age-specific requirements have to be met:

Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution.

Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago.

* Women must not be breastfeeding.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving durvalumab and who are sexually active with WOCBP must be willing to adhere to contraception for a period of 7 month post treatment completion.
* Sexually active men receiving durvalumab must use a condom, even if vasectomized, to prevent delivery of the drug via seminal fluid.

Exclusion Criteria:

* Study participants with squamous cell carcinoma of the esophagus
* Prior treatment with chemotherapy, targeted therapy or radiotherapy for treatment of advanced cancer disease less than 5 years
* Enrollment is possible for patients with:

  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Any other serious or uncontrolled medical disorder, active infections, physical exam findings, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a study participant's ability to comply with the study requirements, substantially increase risk to the study participant, or impact the interpretability or study results
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

Patients with vitiligo or alopecia Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement Any chronic skin condition that does not require systemic therapy Patients without active autoimmune or inflammatory disease in the last 5 years may be included but only after consultation with study physician Patients with celiac disease controlled by diet alone. Inhaled or topical steroids and adrenal replacement steroid doses > 10mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.

* History of active primary immunodeficiency
* History of any allogenic organ transplantation with currently intake of immune suppressive treatment
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity. FEV 1 < 75%
* Patients has known current symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Prisoners or study participants who are involuntarily incarcerated
* Pregnancy or breastfeeding females
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.
* Allergies and Adverse Drug Reaction:

History of allergy to study drug components History of severe hypersensitivity reaction to any monoclonal antibody

• Current treatment within another therapeutic clinical trial with experimental and not approved drugs and treatment combinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Safety and efficacy (measured by an increase of pathological complete response rate) | Calculated once at the end of study (24 months after the end of treatment)
  The primary objective is to evaluate safety and efficacy (measured by an increase of pathological complete response rate from 20% to 35%) of the fully human monoclonal IgG1 antibody durvalumab targeting the programmed death-ligand 1 (PD-L1) in combination with neoadjuvant radiochemotherapy, followed by surgery for locally advanced esophageal cancer and cancer of the gastric esophageal junction (GEJ).

SECONDARY OUTCOMES:
Determination of Best Objective Response (BOR) as defined by RECIST 1.1 and iRECIST criteria after neoadjuvant treatment | Determined once after neoadjuvant treatment (up to 12 weeks after study start)
  To determine the Best Objective Response (BOR) as defined by RECIST 1.1 and iRECIST criteria after neoadjuvant treatment
Determination of Progression Free Survival (PFS) in durvalumab vs. durvalumab + tremelimumab adjuvant treatment | Until 24 months after the end of treatment
  To determine Progression Free Survival (PFS) in durvalumab vs. durvalumab + tremelimumab adjuvant treatment.
  PFS is defined as PFS from treatment start to first detection of disease progression.
Determination of Disease Free Survival (DFS) in durvalumab vs. durvalumab + tremelimumab adjuvant treatment | Until 24 months after the end of treatment
  To determine Disease Free Survival (DFS) in durvalumab vs. durvalumab + tremelimumab adjuvant treatment.
  DFS is defined as DFS from time of surgery to first detection of disease progression.
Determination of Overall Survival (OS) in durvalumab vs. durvalumab + tremelimumab adjuvant treatment | From the study start until the date of death, assessed up to 240 months
  To determine Overall Survival (OS) in durvalumab vs. durvalumab + tremelimumab adjuvant treatment.
  OS is defined as OS from treatment start to death.
Assessment of the subject's esophageal-cancer-related quality of life using the Functional Assessment of Cancer Therapy-Esophageal (FACT-E) questionnaire | Until 24 months after the end of treatment
  To assess the subject's esophageal-cancer-related quality of life using the Functional Assessment of Cancer Therapy-Esophageal (FACT-E) questionnaire.
  The questionnaire will be done by interview administration at screening, visit 5 during neoadjuvant treatment, before surgery, after randomization before start of adjuvant treatment and after then every 12 weeks at the time of tumor staging also in the follow-up phase.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zander, Prof. Dr. med, Principal Investigator — University of Cologne
Locations (2):
- Germany (2):
  - University of Cologne, Cologne
  - Klinikum der Universität München, München

IPD SHARING:
Plan to Share IPD: No